CLINICAL TRIAL: NCT04370587
Title: A Phase 1/2a, Open-Label, Dose Escalation and Expansion Study of the Safety and Tolerability of T3011 Administered Via Intratumoral Injection as a Single Agent and in Combination With Intravenous Pembrolizumab in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Study of Intratumoral MVR-T3011 (T3011) Given as a Single Agent and in Combination With Intravenous Pembrolizumab in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTIV1708
Record Dates: First submitted 2020-04-14; First posted 2020-05-01 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; Melanoma; HNSCC; Sarcoma; Squamous Cell Carcinoma; NSCLC
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Sarcoma; Carcinoma, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1 (Experimental): T3011 single agent dose escalation in participants with solid tumors
  Interventions: Biological: T3011
- Phase 2a Part 1 Arm A (Experimental): RP2D T3011 single agent in participants with melanoma
  Interventions: Biological: T3011
- Phase 2a Part 1 Arm B (Experimental): RP2D T3011 single agent in participants with other solid tumors
  Interventions: Biological: T3011
- Phase 2a Part 2 Arm C (Experimental): RP2D T3011 + pembrolizumab in participants with NSCLC
  Interventions: Combination Product: T3011 + pembrolizumab
- Rollover Arm (Experimental): RP2D T3011 + pembrolizumab in participants who have progressed on T3011 single agent
  Interventions: Combination Product: T3011 + pembrolizumab

INTERVENTIONS:
Biological: T3011 — T3011 will be administered up to 4mL as an intratumoral injection given Q2W.
  Arms: Phase 1; Phase 2a Part 1 Arm A; Phase 2a Part 1 Arm B
Combination Product: T3011 + pembrolizumab — T3011 will be administered up to 4mL as an intratumoral injection in combination with intravenous pembrolizumab given Q3W.
  Arms: Phase 2a Part 2 Arm C; Rollover Arm

SUMMARY:
This is a Phase 1/2a, open-label, study to evaluate the safety and preliminary efficacy of intratumoral T3011 given alone and in combination with intravenous pembrolizumab in partients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, first-in-human study of T3011 given via intratumoral (IT) injection as a single agent and in combination with IV pembrolizumab in participants with advanced or metastatic solid tumors. The Phase 1 portion of the study is a single agent dose escalation which will use a 3+3 design to evaluate escalating doses of T3011. Total enrollment will depend on the toxicities and/or activity observed, with approximately 15 to 30 evaluable participants enrolled. Once the RP2D is established Phase 2a Part 1 will enroll approximately 10 participants with locally recurrent or metastatic melanoma (in Arm A) 23 to 53 participants with HNSCC in Arm B, 40 to 80 participants with sarcoma in Arm C and 10 participants with cSCC in Arm D. During Phase 2a Part 1 the safety, tolerability, and preliminary efficacy of T3011 as a single agent will be evaluated. Phase 2a Part 2 will enroll in parallel to Phase 2a Part 1 once the RP2D is established. The safety, tolerability, and preliminary efficacy of IT T3011 given in combination with IV pembrolizumab will be evaluated in 15 participants with histologically or pathologically confirmed metastatic NSCLC (Arm E). A rollover arm is also included in this study to allow participants who have documented progression on T3011 alone to receive T3011 in combination with pembrolizumab if considered eligible.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18 years or older.
2. Disease progression after standard of care (SOC) therapy or in the opinion of
3. The Investigator unlikely to benefit from SOC therapy. Inclusion Diagnosis Phase 1 - Histologically or pathologically confirmed locally recurrent or metastatic advanced malignancy.

   Phase 2a Part 1 i. Arm A - locally recurrent or metastatic melanoma. Participants must have received no more than 3 prior regimens for advanced or metastatic disease.

   ii. Arm B - locally recurrent or metastatic HNSCC. It must also meet the following criteria: 1) Disease progression to platinum-containing chemotherapy; 2) Failure to anti-PD-1/PDL1 blockade after receiving at least 2 doses alone or in combination.

   iii. Arm C - Sarcoma. Participants must have received no more than three lines of prior anti-cancer therapies.

   iv. Arm D - locally recurrent or metastatic cSCC. Participants must have received no more than 3 prior regimens for advanced or metastatic disease.

   Phase 2a Part 2 i.v. Arm E - Histologically or pathologically confirmed NSCLC that is advanced or recurrent, without EGFR mutation or ALK rearrangement. Participants must have received at least one line but no more than three lines of prior anti-cancer therapies.
4. Measurable disease per RECIST version 1.1.
5. Must have at least 1 tumor lesion that is accessible for IT injection of T3011 in the opinion of the investigator.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. Life expectancy > 12 weeks.
8. Demonstrate adequate organ function as defined by acceptable laboratory testing results.
9. Women of child-bearing potential (WCBP) and men must agree to use adequate contraception prior to study entry, while on study treatment, and for six months after receiving last dose of T3011. WCBP must have a negative serum pregnancy test prior to W1D1.
10. Last dose of previous anticancer therapy ≥ 21 days, radiotherapy > 21 days, or surgical intervention > 21 days prior to the first dose of T3011.
11. Recovered from all prior anticancer therapy toxicities.
12. Willingness to provide fresh tumor biopsy specimens as specified in the Schedule of Assessments.
13. Capable of understanding and complying with protocol requirements.
14. Signed and dated institutional review board/independent ethics committee-approved informed consent form before any protocol-directed screening procedures are performed.

Key Exclusion Criteria:

1. Have only uninjectable tumors..
2. Patients with injectable tumors impinging upon major airways or blood vessels.
3. HNSCC only: Prior re-irradiation field containing carotid artery.
4. Greater than 3 distant metastatic lymph node regions and/or metastatic lesions or the largest distant metastases with a diameter of more than 3 cm (non-sarcoma)/5 cm (sarcoma) unless the lesion is to be injected.
5. Prior treatment with another OV (including T-VEC), tumor vaccines, cellular therapy or gene therapy.
6. Prior intolerance to anti-PD-(L)1 monoclonal antibody or history of immunotherapy related non-infectious pneumonitis/interstitial lung disease.
7. Prior treatment with anti-PD-(L)1 monoclonal antibody in combination with IL-12.
8. Requires continued concurrent therapy with any drug active against HSV.
9. Live vaccines, attenuated vaccines within 4 weeks prior to initiation of study treatment (participants vaccinated with inactivated vaccines can be enrolled.
10. Primary or acquired immunodeficient states.
11. Pregnant or lactating.
12. Prior organ transplantation.
13. Active hepatitis B virus, hepatitis C virus, and HIV infection or a positive serological test at Screening within 14 days of dosing with T3011.
14. Active autoimmune disease or medical conditions requiring chronic steroid or immunosuppressive therapy within 4 weeks prior to first administration of study treatment.
15. History of or current central nervous system metastases.
16. History of seizure disorders within 6 months of Screening.
17. Active oral or skin herpes lesion at Screening.
18. Active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids.
19. Congestive heart failure, active coronary artery disease, unevaluated new onset angina within 3 months or unstable angina, or clinically significant cardiac arrhythmias.
20. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody.

18. Active infection with SARS-CoV-2 virus. 21. Participants with moderate to large amount of pleural effusion, ascites or pericardial effusion who need drug or medical intervention.

22. Other systemic conditions or organ abnormalities that, in the opinion of the investigator, may interfere with the conduct and/or interpretation of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of escalating doses T3011 | Up to 2 years from first dose of T3011
  Number of participants in dose escalating cohorts with dose limiting toxicities (DLTs), treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities.
To determine the dose(s) of T3011 to be examined in Phase 2a | Through the first two T3011 injections (approximately 28 days)
  Incidence of DLTs
Safety and tolerability of T3011 dose(s) selected from Phase 1 in disease specific cohorts | Up to 2 years from first dose of T3011
  Number of participants with treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities.
Characterize the safety and tolerability of T3011 in combination with pembrolizumab | Up to 2 years from first dose of T3011
  Number of participants with treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities.
Characterize the safety and tolerability of T3011 in combination with pembrolizumab in participants who progress on T3011 alone | Up to 2 years from first dose of T3011
  Number of participants with treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years from first dose of T3011
  ORR is defined as the proportion of participants who have a partial response (PR) or complete response (CR) to intervention, based on assessments by RECIST v1.1 and iRECIST.
Disease control rate (DCR) | Up to 2 years from first dose of T3011
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) based on assessments by RECIST v1.1 and iRECIST.
Duration of response (DOR) | Up to 2 years from first dose of T3011
  DOR is defined as the time from the first met CR or PR until disease progression or death due to any cause, whichever occurs first.
Durable response (DR) | Up to 2 years from first dose of T3011
  DR is defined as objective response (CR or PR) according to RECIST v1.1 and iRECIST.
Progression-free survival (PFS) | Up to 2 years from first dose of T3011
  PFS is defined as the time from enrollment to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first per RECIST v1.1 and iRECIST.
Overall Survival (OS) | Up to 1 year after last dose of T3011
  OS is defined as the time from enrollment to death from any cause.
Presence of neutralizing antibodies of anti-PD-1 antibody for antidrug antibodies (ADAs) development | Up to 2 years from first dose of T3011
  To evaluate the immunogenicity of anti-PD-1 antibody expressed by T3011 given as single agent and in combination with pembrolizumab post injection.
Presence and frequency of T3011 in injection site swab, saliva, and urine | Up to 2 years from first dose of T3011
  To evaluate the virus shedding of T3011 following intratumoral injection

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (3):
  - Southern Oncology, Bedford Park
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston
  - The Alfred, Melbourne

IPD SHARING:
Plan to Share IPD: No